CLINICAL TRIAL: NCT04008563
Title: Bariatric Surgery for Fertility-Sparing Treatment of Atypical Hyperplasia and Grade 1 Cancer of the Endometrium
Acronym: B-FiERCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-5487
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer; Atypical Hyperplasia; Bariatric Surgery Candidate
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Intervention Group: Bariatric Surgery and Progestin Intrauterine Device (pIUD) Non-Intervention Group: Progestin Intrauterine Device (pIUD) alone
  Participants who consent will be randomized in a 1:1 allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric Surgery and Progestin Intrauterine Device (Experimental): This group will receive a progestin intrauterine device and be offered to undergo bariatric surgery.
  Interventions: Procedure: Bariatric Surgery
- Progestin Intrauterine Device Alone (No Intervention): This group will receive a progestin intrauterine device alone.

INTERVENTIONS:
Procedure: Bariatric Surgery — Patients who are randomized to the intervention group will receive a progestin intrauterine device and be referred for bariatric service to undergo bariatric surgery within 3 months of their study consent.
  Arms: Bariatric Surgery and Progestin Intrauterine Device

SUMMARY:
A growing population of young women with obesity are developing atypical hyperplasia (pre-cancer) and endometrial cancer. Progestin is the standard treatment for women who wish to preserve fertility, but this approach does not address the underlying cause of endometrial cancer/atypical hyperplasia (obesity); thus response rates are low and recurrence rates are high. Significant weight loss by bariatric surgery, in combination with progestin therapy may result in greater and more durable response rates.

DETAILED DESCRIPTION:
The incidence of endometrial cancer is increasing at an alarming rate (2.6% per year). This trend parallels the rising rate of obesity, the most significant increasing risk factor for endometrial cancer. Young women with obesity and endometrial cancer or atypical hyperplasia who want to maintain their fertility and thus avoid hysterectomy are treated with progestin therapy, such as progestin intra-uterine device (pIUD). However, the pIUD achieves cancer regression in only 50-70% of women, and over 50% of initial responders will develop recurrence within two years. The effectiveness of the pIUD may be improved if the driver of endometrial cancer (obesity) was simultaneously addressed. Multiple epidemiologic studies have demonstrated that bariatric surgery reduces the risk of developing endometrial cancer. Our research aims to answer the question: "Is bariatric surgery in addition to the pIUD a feasible and acceptable option for young women with endometrial cancer/atypical hyperplasia who wish to maintain their childbearing potential compared to standard treatment of pIUD alone?

This is a pilot randomized controlled trial to assess the feasibility of a full-scale randomized controlled trial. Eligible women will be identified and consented over a 21-month period, and participants will be randomized to bariatric surgery plus standard pIUD (intervention group) or to standard pIUD alone (non-intervention group) in a 1:1 fashion.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35
* Diagnosis of grade 1 endometrioid endometrial cancer or complex atypical hyperplasia
* Clinical stage 1 disease - no evidence of metastatic disease beyond the uterus by imaging performed (MRI, CT)
* ECOG status <2
* Desire for fertility preservation
* No contraindications to progestin intrauterine device (IUD)
* Have signed an approved informed consent form

Exclusion Criteria:

* Evidence of myometrial invasion or extra-uterine disease on imaging
* High grade or p53 endometrial cancer
* History of other malignancies, except if curatively treated with no evidence of disease for > 5 years
* Previous major upper abdominal surgery (ex. previous bariatric surgery, splenectomy, partial gastrectomy, liver resection, bowel resection). Appendectomy, cholecystectomy, hernia repair, and caesarean section are acceptable procedures for inclusion.
* Current use of weight loss medication. NB: patients taking glucagon-like peptide 1 (GLP-1) agonists (e.g., OZEMPIC) for the treatment of diabetes will not be excluded.
* Contraindications to sleeve gastrectomy
* Medical co-morbidity with end-organ dysfunction
* Unable to understand and participate in the informed consent process
* Currently pregnant
* Active smoking in ≤6 months
* Active substance use disorder
* Current untreated or severe psychiatric issue

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Year 5
  To determine the proportion of eligible women who agree to participate in the study (recruitment rate). The primary outcome will be met and a full scale randomized controlled trial to assess efficacy will be conducted if ≥ 40% recruitment rate is achieved. Patients' reasons for participation or non-participation will be recorded.

SECONDARY OUTCOMES:
Completion of Bariatric Surgery | Year 5
  Proportion of patients who complete bariatric surgery within 3-4 months (-2/+ 4 weeks) of randomization. A rate of >85% will be considered feasible.
Loss to Follow-Up Rate | Year 6
  Loss to follow-up rate, defined as proportion of patients who do not complete 15-month assessment. A loss to follow-up rate of <20% will be considered feasible.
Completion of Patient Reported Outcome Questionnaires | Year 5
  Completion rate of patient reported outcomes that will be used in the full-scale randomized controlled trial. Completion of >80% of patient reported outcomes at baseline will indicate that use of these questionnaires is feasible.
Complete Response Rate | Year 6
  Overall complete response rate (CRR) after treatment with progestin intrauterine device (pIUD). This study is not powered to detect an improvement in CRR in the intervention vs. non-intervention group. However, the proportion of women who obtain a complete response in the pIUD alone group at 15 months will be used as the baseline CRR for this population and will be used to derive a sample size for a full-scale randomized controlled trial. We believe that this will be more accurate than using published data retrospective studies that are not specific to women with obesity. We will also collect the following data: (a) time to complete response, (b) overall recurrence rate, and (c) time to recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Ferguson, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agnew H, Kitson S, Crosbie EJ. Interventions for weight reduction in obesity to improve survival in women with endometrial cancer. Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD012513. doi: 10.1002/14651858.CD012513.pub3. PMID 36971688